CLINICAL TRIAL: NCT02459678
Title: ART Readiness in HIV-infected Pregnant Women: From Formative Qualitative Research to Individual Randomized Trial
Brief Title: ART Readiness in HIV-infected Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-3884
Record Dates: First submitted 2015-05-14; First posted 2015-06-02 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Other): The MOH-recommended approach is opt out HIV testing in pregnancy followed by immediate initiation of ART for HIV-infected pregnant women. ART initiation is accompanied with counseling geared to educate and prepare women to take up and be retained on ART lifelong. Women who do not return for clinical or drug refill visits are traced by phone or in person.
  Interventions: Other: Standard of Care
- Enhanced adherence package (Experimental): The enhanced adherence package will be designed on the basis of the results of formative research. The intervention will support women who are eligible for ART under Option B+.
  Interventions: Behavioral: Enhanced Adherence Package

INTERVENTIONS:
Behavioral: Enhanced Adherence Package — The enhanced adherence package is yet to be designed, but may target all HIV-infected women with methods that are currently reserved only for late clients or clients of unknown status.
  Arms: Enhanced adherence package
Other: Standard of Care — Currently, the standard of care is based on the 2010 national HIV care and treatment guidelines, health care providers are encouraged to use a number of different means to improve ART adherence.
  Arms: Standard of Care

SUMMARY:
This study seeks to evaluate the readiness of HIV-infected pregnant women in Zambia to initiate, adhere to, and be retained in care under the Ministry of Health's Option B+ policy. Under a 3-phased research study the investigators will: (1) conduct formative research regarding readiness to start lifelong ART in the pregnant population; (2) translate the results of formative research into a readiness assessment tool and an enhanced adherence package for pregnant women eligible for Option B+ and (3) conduct an individual randomized trial of the enhanced adherence package.

DETAILED DESCRIPTION:
This is qualitative and quantitative research exploring the issues of patient readiness to initiate lifelong ART among HIV-infected pregnant women, as well as ART adherence and retention in HIV care and treatment during pregnancy and after delivery.

The objectives of Phase 1 of the study are as follows:

* To identify common themes about patient readiness for ART initiation in the days and weeks following ART eligibility in the context of pregnancy
* To learn about strategies that HIV-infected women and partners of reproductive-age women believe will assist with daily adherence to triple-drug ART and retention in care during pregnancy and after delivery

The objectives of Phase 2 of the study are as follows:

* To develop a screening instrument for assessing readiness of ART initiation during pregnancy
* To pilot the ART readiness assessment tool and evaluate its acceptability and feasibility through qualitative research
* To design a combination intervention that systematically addresses barriers to patient readiness and in so doing, may shorten time from HIV diagnosis to ART initiation and increase rates of ART adherence and retention in care in the short term

The objectives of Phase 3 of the study are as follows:

* To evaluate an enhanced adherence package for improving timely ART initiation and retention in care, defined by attending follow-up ART visit(s), at 30 days after ART eligibility and by maternal HIV viral levels at time of delivery
* To determine the accuracy of the screening instrument in predicting ART readiness by looking at early ART adherence and retention
* To obtain early data about virologic response in pregnancy and postnatal period among HIV-infected women on Option B+
* To obtain data about 6-week and 6-month MTCT rates of HIV among HIV-infected women on Option B+
* To obtain data about renal function in pregnancy and postnatal period among HIV-infected women on Option B+, given that tenofovir is first-line in Zambia

ELIGIBILITY:
The criteria vary by study phase as follows:

Phase 1

Inclusion Criteria:

* HIV-infected pregnant women not yet on ART OR
* HIV-infected pregnant or postnatal women on ART OR
* Partners of women who were recently or are currently pregnant

Exclusion Criteria:

* Less than 18 years old
* Known history of mental illness

Phase 2

Inclusion Criteria:

* HIV-infected pregnant or postnatal women on ART who piloted tested the readiness assessment tool OR
* Health care workers involved in provision of PMTCT and/or ART services at health facility who have pilot tested the readiness assessment tool

Phase 3

Inclusion Criteria:

* Pregnant
* HIV-infected
* Never previously initiated or was on ART for her own health
* Able to provide informed consent
* Willing to undergo all study tests and procedures and be followed until 6 months post-partum

Exclusion criteria:

* Less than 18 years old
* Known intrauterine fetal demise
* Known history of mental illness
* Does not intend to receive antenatal care, labour and delivery care, and postnatal care at the government health facilities of Lusaka District

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Proportion of women who both initiate ART and are retained in care | Within 30 days of eligibility to begin ART under Option B+ policy
  ART eligibility in the setting of Option B+ will generally be either the date of HIV diagnosis for pregnant women newly diagnosed with HIV infection during their antenatal care visit or the date of their first antenatal care visit for known HIV-infected pregnant women who are not already on ART
HIV virologic suppression at time of delivery | Time of delivery
  Outcome of virologic suppression at delivery will be analyzed for differences between the SOC arm and intervention arm.

SECONDARY OUTCOMES:
Time from ART eligibility to ART initiation | Time from ART eligibility to initiation from enrollment until 6 months post-partum
HIV transmission from mother to infant | At 6 weeks and 6 months of life

CONTACTS AND LOCATIONS:
Overall Officials: Mwangelwa Mubiana, MBChB, Principal Investigator — Centre for Infectious Disease Research in Zambia; Benjamin Chi, MD, Principal Investigator — University of North Carolina, Chapel Hill; Michael J Vinikoor, MD, Study Director — Centre for Infectious Disease Research in Zambia
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

REFERENCES:
- [Background] Millennium Development Goals Progress Report. 2011, Ministry of Finance and National Planning, UNDP: Lusaka.
- [Background] National HIV/AIDS/STIs/TB Council, 2009 HIV Epidemiological Projections Report. 2009: Zambia.
- [Background] Republic of Zambia Ministry of Health, National Protocol Guidelines Integrated Prevention of Mother-to-Child Transmission of HIV, Directorate of Public Health and Research, Editor. 2010, Ministry of Health: Lusaka, Zambia.
- [Background] Government of the Republic of Zambia, National Protocol Guidelines Integrated Prevention of Mother-to-Child Transmission of HIV/AIDS, M.o. Health, Editor. 2008: Lusaka.
- [Background] Antiretroviral Drugs for Treating Pregnant Women and Preventing HIV Infection in Infants: Recommendations for a Public Health Approach: 2010 Version. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK304944/ PMID 26180894
- [Background] Centers for Disease Control and Prevention (CDC). Impact of an innovative approach to prevent mother-to-child transmission of HIV--Malawi, July 2011-September 2012. MMWR Morb Mortal Wkly Rep. 2013 Mar 1;62(8):148-51. PMID 23446514
- [Background] Government of the Republic of Zambia, Lifelong Antiretroviral Drugs (ARV's) for all HIV positive Pregnant Women in Zambia, M.o. Health, Editor. 2013: Lusaka.
- [Background] Government of the Republic of Zambia, Adult and Adolescent Antiretroviral Therapy Protocols, M.o. Health, Editor. 2010: Lusaka.
- [Background] Shaffer N, Abrams EJ, Becquet R. Option B+ for prevention of mother-to-child transmission of HIV in resource-constrained settings: great promise but some early caution. AIDS. 2014 Feb 20;28(4):599-601. doi: 10.1097/QAD.0000000000000144. No abstract available. PMID 24469000
- [Background] Tenthani L, Haas AD, Tweya H, Jahn A, van Oosterhout JJ, Chimbwandira F, Chirwa Z, Ng'ambi W, Bakali A, Phiri S, Myer L, Valeri F, Zwahlen M, Wandeler G, Keiser O. Retention in care under universal antiretroviral therapy for HIV-infected pregnant and breastfeeding women ('Option B+') in Malawi. AIDS. 2014 Feb 20;28(4):589-598. doi: 10.1097/QAD.0000000000000143. PMID 24468999
- [Background] UNAIDS. HIV and AIDS estimates 2009. [cited 2011 April 11]; Available from: http://www.unaids.org/en/regionscountries/countries/zambia/.
- [Background] Zambia National HIV/AIDS/STI/TB Council, Zambia HIV Prevention Response and Modes of Transmission Analysis. 2009.
- [Background] Mazimba C, C.W., , Kaseba C, Chi B, HIV-related maternal mortality in Lusaka, Zambia: 1993-2004, in 3rd IAS Conference on HIV Pathogenesis and Treatment: Rio de Janeiro, Brazil.
- [Background] Moodley J, Pattinson RC, Baxter C, Sibeko S, Abdool Karim Q. Strengthening HIV services for pregnant women: an opportunity to reduce maternal mortality rates in Southern Africa/sub-Saharan Africa. BJOG. 2011 Jan;118(2):219-25. doi: 10.1111/j.1471-0528.2010.02726.x. Epub 2010 Sep 24. PMID 21159120
- [Background] McIntyre J. Maternal health and HIV. Reprod Health Matters. 2005 May;13(25):129-35. doi: 10.1016/s0968-8080(05)25184-4. PMID 16035606
- [Background] Kuhn L, Aldrovandi GM, Sinkala M, Kankasa C, Semrau K, Kasonde P, Mwiya M, Tsai WY, Thea DM; Zambia Exclusive Breastfeeding Study (ZEBS). Differential effects of early weaning for HIV-free survival of children born to HIV-infected mothers by severity of maternal disease. PLoS One. 2009 Jun 26;4(6):e6059. doi: 10.1371/journal.pone.0006059. PMID 19557167
- [Background] Kuhn L, Aldrovandi GM, Sinkala M, Kankasa C, Mwiya M, Thea DM. Potential impact of new WHO criteria for antiretroviral treatment for prevention of mother-to- child HIV transmission. AIDS. 2010 Jun 1;24(9):1374-7. PMID 20568677
- [Background] Sewankambo NK, Gray RH, Ahmad S, Serwadda D, Wabwire-Mangen F, Nalugoda F, Kiwanuka N, Lutalo T, Kigozi G, Li C, Meehan MP, Brahmbatt H, Wawer MJ. Mortality associated with HIV infection in rural Rakai District, Uganda. AIDS. 2000 Oct 20;14(15):2391-400. doi: 10.1097/00002030-200010200-00021. PMID 11089628
- [Background] Bicego G, Boerma JT, Ronsmans C. The effect of AIDS on maternal mortality in Malawi and Zimbabwe. AIDS. 2002 May 3;16(7):1078-81. doi: 10.1097/00002030-200205030-00019. No abstract available. PMID 11953479
- [Background] Morgenstern TT, Grimes DE, Grimes RM. Assessment of readiness to initiate antiretroviral therapy. HIV Clin Trials. 2002 Mar-Apr;3(2):168-72. doi: 10.1310/T6Y6-BRCW-AR7A-WVA3. PMID 11976996
- [Background] Nachega JB, Uthman OA, Anderson J, Peltzer K, Wampold S, Cotton MF, Mills EJ, Ho YS, Stringer JS, McIntyre JA, Mofenson LM. Adherence to antiretroviral therapy during and after pregnancy in low-income, middle-income, and high-income countries: a systematic review and meta-analysis. AIDS. 2012 Oct 23;26(16):2039-52. doi: 10.1097/QAD.0b013e328359590f. PMID 22951634
- [Background] Weigel R, Hosseinipour MC, Feldacker C, Gareta D, Tweya H, Chiwoko J, Gumulira J, Kalulu M, Mofolo I, Kamanga E, Mwale G, Kadzakumanja A, Jere E, Phiri S. Ensuring HIV-infected pregnant women start antiretroviral treatment: an operational cohort study from Lilongwe, Malawi. Trop Med Int Health. 2012 Jun;17(6):751-9. doi: 10.1111/j.1365-3156.2012.02980.x. Epub 2012 Apr 5. PMID 22487553
- [Background] Wagner GJ, Goggin K, Remien RH, Rosen MI, Simoni J, Bangsberg DR, Liu H; MACH14 Investigators. A closer look at depression and its relationship to HIV antiretroviral adherence. Ann Behav Med. 2011 Dec;42(3):352-60. doi: 10.1007/s12160-011-9295-8. PMID 21818528
- [Background] Balfour L, Kowal J, Silverman A, Tasca GA, Angel JB, Macpherson PA, Garber G, Cooper CL, Cameron DW. A randomized controlled psycho-education intervention trial: Improving psychological readiness for successful HIV medication adherence and reducing depression before initiating HAART. AIDS Care. 2006 Oct;18(7):830-8. doi: 10.1080/09540120500466820. PMID 16971295
- [Background] Tremblay CL, Baril JG, Fletcher D, Kilby D, Macpherson P, Shafran SD, Tyndall MW. Challenges in initiating antiretroviral therapy in 2010. Can J Infect Dis Med Microbiol. 2010 Aug;21 Suppl C(Suppl C):1C-15C. PMID 23365594
- [Background] Fehr JS, Nicca D, Sendi P, Wolf E, Wagels T, Kiss A, Bregenzer T, Vernazza P, Jager H, Spirig R, Battegay M; Swiss HIV Cohort Study. Starting or changing therapy - a prospective study exploring antiretroviral decision-making. Infection. 2005 Aug;33(4):249-56. doi: 10.1007/s15010-005-4141-1. PMID 16091895
- [Background] Wolff B, Mbonye M, Coutinho A, Amuron B, Nkabala R, Jaffar S, Grosskurth H. High levels of psychosocial readiness for ART in an African population at the onset of treatment. SAHARA J. 2009 Dec;6(4):188-94. doi: 10.1080/17290376.2009.9724947. PMID 20485858
- [Background] Macdonell KE, Naar-King S, Murphy DA, Parsons JT, Harper GW. Predictors of medication adherence in high risk youth of color living with HIV. J Pediatr Psychol. 2010 Jul;35(6):593-601. doi: 10.1093/jpepsy/jsp080. Epub 2009 Sep 15. PMID 19755495
- [Background] Tessema B, Biadglegne F, Mulu A, Getachew A, Emmrich F, Sack U. Magnitude and determinants of nonadherence and nonreadiness to highly active antiretroviral therapy among people living with HIV/AIDS in Northwest Ethiopia: a cross-sectional study. AIDS Res Ther. 2010 Jan 14;7:2. doi: 10.1186/1742-6405-7-2. PMID 20180959
- [Background] Central Statistical Office, Demographic Health Survey. 2007: Lusaka.
- [Background] Weiss L, French T, Finkelstein R, Waters M, Mukherjee R, Agins B. HIV-related knowledge and adherence to HAART. AIDS Care. 2003 Oct;15(5):673-9. doi: 10.1080/09540120310001595159. PMID 12959818
- [Background] Johnson MO, Gamarel KE, Dawson Rose C. Changing HIV treatment expectancies: a pilot study. AIDS Care. 2006 Aug;18(6):550-3. doi: 10.1080/09540120500241439. PMID 16831781
- [Background] Pence BW, Ostermann J, Kumar V, Whetten K, Thielman N, Mugavero MJ. The influence of psychosocial characteristics and race/ethnicity on the use, duration, and success of antiretroviral therapy. J Acquir Immune Defic Syndr. 2008 Feb 1;47(2):194-201. doi: 10.1097/QAI.0b013e31815ace7e. PMID 17971712
- [Background] Johnson MO, Dilworth SE, Stephens E, Lum PJ, Neilands TB. Expectancy and readiness-based predictors of treatment uptake among the urban poor living with HIV. J Acquir Immune Defic Syndr. 2011 Dec 15;58(5):469-71. doi: 10.1097/QAI.0b013e3182365671. PMID 21926630
- [Background] Grimes RM, Grimes DE. Patient readiness to adhere to HAART. J Int Assoc Physicians AIDS Care (Chic). 2009 Nov-Dec;8(6):364-6. doi: 10.1177/1545109709351240. PMID 19952288
- [Background] Wagner G, Iguchi M, Schneider S, Scott J, Anderson D. Placebo practice trials: a tool to assess and improve adherence readiness. HIV Clin Trials. 2002 Nov-Dec;3(6):475-81. doi: 10.1310/WQRY-FNUL-VNE1-56XA. PMID 12501131
- [Background] Wagner GJ, Kanouse DE, Koegel P, Sullivan G. Correlates of HIV antiretroviral adherence in persons with serious mental illness. AIDS Care. 2004 May;16(4):501-6. doi: 10.1080/09540120410001683420. PMID 15203417
- [Background] Willey C, Redding C, Stafford J, Garfield F, Geletko S, Flanigan T, Melbourne K, Mitty J, Caro JJ. Stages of change for adherence with medication regimens for chronic disease: development and validation of a measure. Clin Ther. 2000 Jul;22(7):858-71. doi: 10.1016/s0149-2918(00)80058-2. PMID 10945512
- [Background] Konkle-Parker DJ. A motivational intervention to improve adherence to treatment of chronic disease. J Am Acad Nurse Pract. 2001 Feb;13(2):61-8. doi: 10.1111/j.1745-7599.2001.tb00219.x. PMID 11930399
- [Background] Thompson MA, Mugavero MJ, Amico KR, Cargill VA, Chang LW, Gross R, Orrell C, Altice FL, Bangsberg DR, Bartlett JG, Beckwith CG, Dowshen N, Gordon CM, Horn T, Kumar P, Scott JD, Stirratt MJ, Remien RH, Simoni JM, Nachega JB. Guidelines for improving entry into and retention in care and antiretroviral adherence for persons with HIV: evidence-based recommendations from an International Association of Physicians in AIDS Care panel. Ann Intern Med. 2012 Jun 5;156(11):817-33, W-284, W-285, W-286, W-287, W-288, W-289, W-290, W-291, W-292, W-293, W-294. doi: 10.7326/0003-4819-156-11-201206050-00419. Epub 2012 Mar 5. PMID 22393036
- [Background] Balfour L, Tasca GA, Kowal J, Corace K, Cooper CL, Angel JB, Garber G, Macpherson PA, Cameron DW. Development and validation of the HIV Medication Readiness Scale. Assessment. 2007 Dec;14(4):408-16. doi: 10.1177/1073191107304295. PMID 17986658
- [Background] Grimes RM, Grimes DE. Readiness: the state of the science (or the lack thereof). Curr HIV/AIDS Rep. 2010 Nov;7(4):245-52. doi: 10.1007/s11904-010-0056-2. PMID 20714831
- [Background] Fernandez MI, Hosek S, Warren JC, Jacobs RJ, Hernandez N, Martinez J; Adolescent Medicine Trials Network (ATN). Development of an easy to use tool to assess HIV treatment readiness in adolescent clinical care settings. AIDS Care. 2011 Nov;23(11):1492-9. doi: 10.1080/09540121.2011.565020. Epub 2011 Jun 21. PMID 22022853
- [Background] Chi BH, Bolton-Moore C, Holmes CB. Prevention of mother-to-child HIV transmission within the continuum of maternal, newborn, and child health services. Curr Opin HIV AIDS. 2013 Sep;8(5):498-503. doi: 10.1097/COH.0b013e3283637f7a. PMID 23872611
- [Background] Stubbs BA, Micek MA, Pfeiffer JT, Montoya P, Gloyd S. Treatment partners and adherence to HAART in Central Mozambique. AIDS Care. 2009 Nov;21(11):1412-9. doi: 10.1080/09540120902814395. PMID 20024718
- [Background] Cook PF, McCabe MM, Emiliozzi S, Pointer L. Telephone nurse counseling improves HIV medication adherence: an effectiveness study. J Assoc Nurses AIDS Care. 2009 Jul-Aug;20(4):316-25. doi: 10.1016/j.jana.2009.02.008. PMID 19576548
- [Background] Rodrigues R, Shet A, Antony J, Sidney K, Arumugam K, Krishnamurthy S, D'Souza G, DeCosta A. Supporting adherence to antiretroviral therapy with mobile phone reminders: results from a cohort in South India. PLoS One. 2012;7(8):e40723. doi: 10.1371/journal.pone.0040723. Epub 2012 Aug 27. PMID 22952574
- [Background] Seidenberg P, Nicholson S, Schaefer M, Semrau K, Bweupe M, Masese N, Bonawitz R, Chitembo L, Goggin C, Thea DM. Early infant diagnosis of HIV infection in Zambia through mobile phone texting of blood test results. Bull World Health Organ. 2012 May 1;90(5):348-56. doi: 10.2471/BLT.11.100032. PMID 22589568
- [Background] Webster PD, Sibanyoni M, Malekutu D, Mate KS, Venter WD, Barker PM, Moleko W. Using quality improvement to accelerate highly active antiretroviral treatment coverage in South Africa. BMJ Qual Saf. 2012 Apr;21(4):315-24. doi: 10.1136/bmjqs-2011-000381. PMID 22438327
- [Background] Assefa Y, Kiflie A, Tekle B, Mariam DH, Laga M, Van Damme W. Effectiveness and acceptability of delivery of antiretroviral treatment in health centres by health officers and nurses in Ethiopia. J Health Serv Res Policy. 2012 Jan;17(1):24-9. doi: 10.1258/jhsrp.2011.010135. Epub 2011 Nov 17. PMID 22096081
- [Background] Perez F, Aung KD, Ndoro T, Engelsmann B, Dabis F. Participation of traditional birth attendants in prevention of mother-to-child transmission of HIV services in two rural districts in Zimbabwe: a feasibility study. BMC Public Health. 2008 Dec 5;8:401. doi: 10.1186/1471-2458-8-401. PMID 19061506
- [Background] Borghi J, Ensor T, Somanathan A, Lissner C, Mills A; Lancet Maternal Survival Series steering group. Mobilising financial resources for maternal health. Lancet. 2006 Oct 21;368(9545):1457-65. doi: 10.1016/S0140-6736(06)69383-5. PMID 17055948
- [Background] Schmidt JO, Ensor T, Hossain A, Khan S. Vouchers as demand side financing instruments for health care: a review of the Bangladesh maternal voucher scheme. Health Policy. 2010 Jul;96(2):98-107. doi: 10.1016/j.healthpol.2010.01.008. PMID 20138385
- [Background] Ekirapa-Kiracho E, Waiswa P, Rahman MH, Makumbi F, Kiwanuka N, Okui O, Rutebemberwa E, Bua J, Mutebi A, Nalwadda G, Serwadda D, Pariyo GW, Peters DH. Increasing access to institutional deliveries using demand and supply side incentives: early results from a quasi-experimental study. BMC Int Health Hum Rights. 2011 Mar 9;11 Suppl 1(Suppl 1):S11. doi: 10.1186/1472-698X-11-S1-S11. PMID 21410998
- [Background] Kalembo FW, Zgambo M, Mulaga AN, Yukai D, Ahmed NI. Association between male partner involvement and the uptake of prevention of mother-to-child transmission of HIV (PMTCT) interventions in Mwanza district, Malawi: a retrospective cohort study. PLoS One. 2013 Jun 12;8(6):e66517. doi: 10.1371/journal.pone.0066517. Print 2013. PMID 23776683
- [Background] Myer L, Zulliger R, Bekker LG, Abrams E. Systemic delays in the initiation of antiretroviral therapy during pregnancy do not improve outcomes of HIV-positive mothers: a cohort study. BMC Pregnancy Childbirth. 2012 Sep 11;12:94. doi: 10.1186/1471-2393-12-94. PMID 22963318
- [Background] Krueger, R. and M. Casey, Focus Groups: A Practical Guide for Applied Research, 3rd edition. 2000, Thousand Oaks: Sage Publications.
- [Background] Nordqvist O, Sodergard B, Tully MP, Sonnerborg A, Lindblad AK. Assessing and achieving readiness to initiate HIV medication. Patient Educ Couns. 2006 Jul;62(1):21-30. doi: 10.1016/j.pec.2005.09.014. PMID 16766244
- [Background] Bernard, H.R., Research Methods in Anthropology. 1995, Walnut Creek Altamira Press 535.
- [Background] Miles, M. and A. Huberman, Qualitative Data Analysis: An Expanded Sourcebook. 2nd ed. 1994, Thousand Oaks: Sage Publications.
- [Background] Enriquez M, Lackey NR, O'Connor MC, McKinsey DS. Successful adherence after multiple HIV treatment failures. J Adv Nurs. 2004 Feb;45(4):438-46. doi: 10.1046/j.1365-2648.2003.02928.x. PMID 14756838
- [Background] Gerbert B, Bronstone A, Clanon K, Abercrombie P, Bangsberg D. Combination antiretroviral therapy: health care providers confront emerging dilemmas. AIDS Care. 2000 Aug;12(4):409-21. doi: 10.1080/09540120050123819. PMID 11091774
- [Background] Chibwesha CJ, Giganti MJ, Putta N, Chintu N, Mulindwa J, Dorton BJ, Chi BH, Stringer JS, Stringer EM. Optimal time on HAART for prevention of mother-to-child transmission of HIV. J Acquir Immune Defic Syndr. 2011 Oct 1;58(2):224-8. doi: 10.1097/QAI.0b013e318229147e. PMID 21709566
- [Background] European Collaborative Study; Patel D, Cortina-Borja M, Thorne C, Newell ML. Time to undetectable viral load after highly active antiretroviral therapy initiation among HIV-infected pregnant women. Clin Infect Dis. 2007 Jun 15;44(12):1647-56. doi: 10.1086/518284. Epub 2007 May 2. PMID 17516411
- [Background] Naar-King S, Parsons JT, Murphy D, Kolmodin K, Harris DR; ATN 004 Protocol Team. A multisite randomized trial of a motivational intervention targeting multiple risks in youth living with HIV: initial effects on motivation, self-efficacy, and depression. J Adolesc Health. 2010 May;46(5):422-8. doi: 10.1016/j.jadohealth.2009.11.198. Epub 2010 Feb 4. PMID 20413077
- [Derived] Mubiana-Mbewe M, Bosomprah S, Kadota JL, Koyuncu A, Kusanathan T, Mweebo K, Musokotwane K, Mulenga PL, Chi BH, Vinikoor MJ. Effect of Enhanced Adherence Package on Early ART Uptake Among HIV-Positive Pregnant Women in Zambia: An Individual Randomized Controlled Trial. AIDS Behav. 2021 Mar;25(3):992-1000. doi: 10.1007/s10461-020-03060-4. Epub 2020 Oct 8. PMID 33033996
- See also: University of North Carolina website — http://www.unc.edu